CLINICAL TRIAL: NCT02802878
Title: Determining the Effects of the Combined Application of Electrical Stimulation and Volitional Contractions on Muscle Strength and Knee Pain and Function in Women With or at Risk for Knee Osteoarthritis
Brief Title: Combined Application of Electrical Stimulation and Volitional Contractions for Muscle Strengthening and Knee Pain Inhibition (Seated Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Kurume University (Other)
Responsible Party: Principal Investigator, Neil Segal, MD, MS, Professor and Faculty Physiatrist, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003872
Record Dates: First submitted 2016-06-09; First posted 2016-06-16 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hybrid Training (Experimental): The hybrid training system combines the applications of neuromuscular electrical stimulation (NMES) with voluntary contractions (NMES-VC). Training will be performed in a seated position with feet not touching the ground, and will involve each knee flexing and extending alternately. The joint range of motion will be restricted to a 90º arc from approximately 10º to 100º of flexion. Each session will consist of 5 sets of 10 repetitions, 3-second knee flexion and extension contractions on each leg. Sets will be separated by 30-sec rest intervals.
  Electrodes will be placed on the anterior thigh over the motor points of the bilateral vastus medialis and lateralis, and over the medial and lateral hamstrings on the posterior thigh. Electrical stimulation intensity will be set to approximately 40% of 1 repetition maximum (RM). A joint motion sensor will trigger stimulation of the antagonist once it senses the initiation of volitional contraction of the agonist muscle group.
  Interventions: Device: Hybrid Training using Electrodes and Joint Motion Sensors
- Low Intensity Exercise (Active Comparator): 40% 1-repetition maximum isokinetic training with HUMAC NORM in same repetitions/sets as experimental group.
  Interventions: Device: Isokinetic Training with Isokinetic Dynamometer

INTERVENTIONS:
Device: Hybrid Training using Electrodes and Joint Motion Sensors — Electrodes (Sekisui Plastics Co., Tokyo, Japan) will be placed on the anterior thigh over the motor points of the bilateral vastus medialis and lateralis, and on the posterior thigh over the motor points of the medial and lateral hamstrings. Electrical stimulation intensity will be set to approximately 40% of 1 repetition maximum (RM).
  A joint motion sensor (Mutoh Engineering Inc., Tokyo, Japan) will trigger stimulation of the antagonist once it senses the initiation of volitional contraction of the agonist muscle group.
  Arms: Hybrid Training
Device: Isokinetic Training with Isokinetic Dynamometer — Low intensity exercises completed using isokinetic dynamometer (HUMAC NORM, Computer Sports Medicine Inc. (CSMi), Stoughton, MA) in isokinetic mode at approximately 40%1 RM.
  Other Names: Resistance Training
  Arms: Low Intensity Exercise

SUMMARY:
The purpose of this study is to assess the efficacy of a 12-week low-load neuromuscular electrical stimulation with volitional contraction (NMES-VC) training program to improve quadriceps strength and activation, while not adversely affecting knee-related pain, activities of daily living or quality of life in women with knee pain. The primary outcome will be change in maximal isokinetic knee extensor torque.

The investigators will test the following hypotheses. In comparison with low-load (40%) resistance training without electrical stimulation, a 12-week NMES-VC training program will:

Hypothesis 1: Increase maximal isokinetic knee extensor torque

Secondary questions and response variables

Hypothesis 2: Not adversely affect knee pain or quality of life, assessed by the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire

Additional hypotheses in women with risk factors for incident symptomatic or progressive KOA:

1. Determine the extent to which NMES-VC-enhanced low-intensity resistance training increases quadriceps muscle rate of force development
2. Determine the extent to which NMES-VC enhanced low-intensity exercise is tolerated (using numeric rating scale survey "level of pain you experienced during the hybrid training or 40% isokinetic exercise")
3. Determine the extent to which NMES-VC-enhanced low-intensity resistance training increases physical function (20m walk, chair stand)

DETAILED DESCRIPTION:
Arthritis is the most common cause of disability in the United States. Approximately 42.1% of women and 31.2% of men over the age of 60 have knee osteoarthritis (KOA). KOA is associated with pain, quadriceps weakness, swelling, instability, decline of range of motion, physical function, and quality of life (QOL). The presence of KOA significantly decreases QOL, while quadriceps strengthening has the ability to improve QOL. However, one challenge with strengthening is that knee pain influences muscle strength and physical function. Not only quadriceps strengthening but also reduction of knee pain may be necessary to reduce functional limitations from KOA. However, at this time, there is insufficient evidence regarding effective training to not only increase quadriceps strength but also reduce knee pain and improve neural function. Thus, there is a need for interventional studies to build on observational findings to evaluate the relationships of neural function, knee muscle strength, knee pain, and physical function.

The critical barrier to studying whether quadriceps strengthening is protective against worsening physical function is the lack of an effective strengthening program for people at elevated risk for KOA. Factors that place older adults at elevated risk for symptomatic KOA, (e.g. sedentary lifestyle, obesity, knee pain, knee injury or surgery), may also contribute to reduced tolerance of high load quadriceps strengthening programs. If a well-tolerated and effective means of strengthening could be identified, it may also have additional benefits in reducing knee pain, improving physical function and avoiding disability in individuals with or at risk of KOA.

Neuromuscular electrical stimulation (NMES) is widely used to strengthen muscles and improve function in people who cannot exercise at medium-high intensity. For KOA, NMES is effective for enhancing quadriceps strength, knee pain, physical function. Therefore, NMES could contribute to decreased neural inhibition from knee pain and promote muscle function (e.g. muscle strength, power, contraction speed, and co-contraction). Recently, it was reported that the combined application of NMES and volitional contractions (NMES-VC) is effective for making up for a limitation of NMES. NMES-VC could help to improve motor recovery. The results of recent studies suggest that a hybrid training system that utilizes both volitional contractions and NMES simultaneously, might be an effective method that can improve physical function by strengthening muscles and relieving knee pain in people at risk for incident or progressive symptomatic KOA.

This line of research could have a significant positive impact on public health, by leading to the introduction of an inexpensive means of well-tolerated and safe exercise that can be completed in community rehabilitative environments. Successful completion of this initial investigation will enable pursuit of research to determine whether NMES-VC is effective in quadriceps strengthening and pain relief while improving neural function in symptomatic and progressive KOA. Reduction of this primary cause of disability through cost-effective preventive exercise has a high potential to reduce the burden of disease and disablement, thereby improving the quality of life for older adults and significantly reducing the costs to individuals and society.

The specific aim of the proposed research is to assess the efficacy of a twelve-week, efficient and tolerable, low-intensity exercise program with NMES-VC for improving quadriceps strength, knee pain and physical function in women with risk factors for incident symptomatic or progressive KOA. This specific aim will be achieved through a randomized, controlled trial, comparing low intensity exercise with and without NMES-VC. This research is novel in that it will be the first to use a low load regimen that will minimize the potential for adverse loading on the knee joint while still having a high likelihood to lead to clinically meaningful strength gains, pain relief and physical function improvement in older adults at elevated risk for symptomatic or progressive KOA.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age 40-85 years
3. One or more of the following:

   1. Knee symptoms (pain, aching, or stiffness) on most of the last 30 days; categorically defined, so all severity of symptoms ok, but must have knee symptoms on most days
   2. History of knee injury or surgery
   3. Body Mass Index (BMI) greater than or equal to 25 kg/m2
4. BMI less than 45 kg/m2

Exclusion Criteria:

1. Knee injection within 6 weeks prior to the study
2. Resistance training at any time in the last 3 months prior to the study
3. Bilateral knee replacement
4. Lower limb amputation
5. Lower limb surgery in the last 6 months that affects walking ability or ability to exercise
6. Back, hip or knee problems that affect walking ability or ability to exercise
7. Unable to walk without a cane or walker
8. Inflammatory joint or muscle disease such as rheumatoid or psoriatic arthritis or polymyalgia rheumatica
9. Multiple sclerosis or other neurodegenerative disorder
10. Known neuropathy
11. Self-report of Diabetes
12. Currently being treated for cancer or having untreated cancer
13. Terminal illness (cannot be cured or adequately treated and there is a reasonable expectation of death in the near future)
14. Peripheral Vascular Disease
15. History of myocardial infarction or stroke in the last year
16. Chest pain during exercise or at rest
17. Use of supplemental oxygen
18. Inability to follow protocol (e.g. lack of ability to attend visits or understand instructions)
19. Staff concern for participant health (such as history of dizziness/faintness or current restrictions on activity)
20. Unable to attend 12 or more sessions during the study
21. Implanted cardiac pacemaker, spinal cord stimulator, baclofen or morphine pump or other implanted electrical device.
22. Dermatitis or skin sensitivity.
23. Pregnancy

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12-14 (Actual); Study Completion 2016-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Segal, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence and most common causes of disability among adults--United States, 2005. MMWR Morb Mortal Wkly Rep. 2009 May 1;58(16):421-6. PMID 19407734
- [Background] Dillon CF, Rasch EK, Gu Q, Hirsch R. Prevalence of knee osteoarthritis in the United States: arthritis data from the Third National Health and Nutrition Examination Survey 1991-94. J Rheumatol. 2006 Nov;33(11):2271-9. Epub 2006 Oct 1. PMID 17013996
- [Background] Segal NA, Glass NA, Felson DT, Hurley M, Yang M, Nevitt M, Lewis CE, Torner JC. Effect of quadriceps strength and proprioception on risk for knee osteoarthritis. Med Sci Sports Exerc. 2010 Nov;42(11):2081-8. doi: 10.1249/MSS.0b013e3181dd902e. PMID 20351594
- [Background] Segal NA, Torner JC, Felson D, Niu J, Sharma L, Lewis CE, Nevitt M. Effect of thigh strength on incident radiographic and symptomatic knee osteoarthritis in a longitudinal cohort. Arthritis Rheum. 2009 Sep 15;61(9):1210-7. doi: 10.1002/art.24541. PMID 19714608
- [Background] van Dijk GM, Dekker J, Veenhof C, van den Ende CH; Carpa Study Group. Course of functional status and pain in osteoarthritis of the hip or knee: a systematic review of the literature. Arthritis Rheum. 2006 Oct 15;55(5):779-85. doi: 10.1002/art.22244. PMID 17013827
- [Background] McAlindon TE, Cooper C, Kirwan JR, Dieppe PA. Determinants of disability in osteoarthritis of the knee. Ann Rheum Dis. 1993 Apr;52(4):258-62. doi: 10.1136/ard.52.4.258. PMID 8484690
- [Background] Palmieri RM, Tom JA, Edwards JE, Weltman A, Saliba EN, Mistry DJ, Ingersoll CD. Arthrogenic muscle response induced by an experimental knee joint effusion is mediated by pre- and post-synaptic spinal mechanisms. J Electromyogr Kinesiol. 2004 Dec;14(6):631-40. doi: 10.1016/j.jelekin.2004.06.002. PMID 15491837
- [Background] Heroux ME, Tremblay F. Corticomotor excitability associated with unilateral knee dysfunction secondary to anterior cruciate ligament injury. Knee Surg Sports Traumatol Arthrosc. 2006 Sep;14(9):823-33. doi: 10.1007/s00167-006-0063-4. Epub 2006 Feb 25. PMID 16502299
- [Background] Palmieri RM, Ingersoll CD, Edwards JE, Hoffman MA, Stone MB, Babington JP, Cordova ML, Krause BA. Arthrogenic muscle inhibition is not present in the limb contralateral to a simulated knee joint effusion. Am J Phys Med Rehabil. 2003 Dec;82(12):910-6. doi: 10.1097/01.PHM.0000098045.04883.02. PMID 14627927
- [Background] Muraki S, Akune T, Oka H, Ishimoto Y, Nagata K, Yoshida M, Tokimura F, Nakamura K, Kawaguchi H, Yoshimura N. Incidence and risk factors for radiographic knee osteoarthritis and knee pain in Japanese men and women: a longitudinal population-based cohort study. Arthritis Rheum. 2012 May;64(5):1447-56. doi: 10.1002/art.33508. PMID 22135156
- [Background] Slemenda C, Brandt KD, Heilman DK, Mazzuca S, Braunstein EM, Katz BP, Wolinsky FD. Quadriceps weakness and osteoarthritis of the knee. Ann Intern Med. 1997 Jul 15;127(2):97-104. doi: 10.7326/0003-4819-127-2-199707150-00001. PMID 9230035
- [Background] Aguiar GC, Do Nascimento MR, De Miranda AS, Rocha NP, Teixeira AL, Scalzo PL. Effects of an exercise therapy protocol on inflammatory markers, perception of pain, and physical performance in individuals with knee osteoarthritis. Rheumatol Int. 2015 Mar;35(3):525-31. doi: 10.1007/s00296-014-3148-2. Epub 2014 Oct 10. PMID 25300730
- [Background] Vincent KR, Vincent HK. Resistance exercise for knee osteoarthritis. PM R. 2012 May;4(5 Suppl):S45-52. doi: 10.1016/j.pmrj.2012.01.019. PMID 22632702
- [Background] Glass NA, Torner JC, Frey Law LA, Wang K, Yang T, Nevitt MC, Felson DT, Lewis CE, Segal NA. The relationship between quadriceps muscle weakness and worsening of knee pain in the MOST cohort: a 5-year longitudinal study. Osteoarthritis Cartilage. 2013 Sep;21(9):1154-9. doi: 10.1016/j.joca.2013.05.016. PMID 23973125
- [Background] Sattler M, Dannhauer T, Hudelmaier M, Wirth W, Sanger AM, Kwoh CK, Hunter DJ, Eckstein F; OAI investigators. Side differences of thigh muscle cross-sectional areas and maximal isometric muscle force in bilateral knees with the same radiographic disease stage, but unilateral frequent pain - data from the osteoarthritis initiative. Osteoarthritis Cartilage. 2012 Jun;20(6):532-40. doi: 10.1016/j.joca.2012.02.635. Epub 2012 Mar 3. PMID 22395037
- [Background] Apkarian AV, Bushnell MC, Treede RD, Zubieta JK. Human brain mechanisms of pain perception and regulation in health and disease. Eur J Pain. 2005 Aug;9(4):463-84. doi: 10.1016/j.ejpain.2004.11.001. Epub 2005 Jan 21. PMID 15979027
- [Background] Campos GE, Luecke TJ, Wendeln HK, Toma K, Hagerman FC, Murray TF, Ragg KE, Ratamess NA, Kraemer WJ, Staron RS. Muscular adaptations in response to three different resistance-training regimens: specificity of repetition maximum training zones. Eur J Appl Physiol. 2002 Nov;88(1-2):50-60. doi: 10.1007/s00421-002-0681-6. Epub 2002 Aug 15. PMID 12436270
- [Background] Hurley MV, Scott DL. Improvements in quadriceps sensorimotor function and disability of patients with knee osteoarthritis following a clinically practicable exercise regime. Br J Rheumatol. 1998 Nov;37(11):1181-7. doi: 10.1093/rheumatology/37.11.1181. PMID 9851266
- [Background] Balogun JA, Onilari OO, Akeju OA, Marzouk DK. High voltage electrical stimulation in the augmentation of muscle strength: effects of pulse frequency. Arch Phys Med Rehabil. 1993 Sep;74(9):910-6. PMID 8379835
- [Background] Delitto A, Rose SJ, McKowen JM, Lehman RC, Thomas JA, Shively RA. Electrical stimulation versus voluntary exercise in strengthening thigh musculature after anterior cruciate ligament surgery. Phys Ther. 1988 May;68(5):660-3. doi: 10.1093/ptj/68.5.660. PMID 3258994
- [Background] Kagaya H, Shimada Y, Ebata K, Sato M, Sato K, Yukawa T, Obinata G. Restoration and analysis of standing-up in complete paraplegia utilizing functional electrical stimulation. Arch Phys Med Rehabil. 1995 Sep;76(9):876-81. doi: 10.1016/s0003-9993(95)80556-7. PMID 7668962
- [Background] Snyder-Mackler L, Delitto A, Bailey SL, Stralka SW. Strength of the quadriceps femoris muscle and functional recovery after reconstruction of the anterior cruciate ligament. A prospective, randomized clinical trial of electrical stimulation. J Bone Joint Surg Am. 1995 Aug;77(8):1166-73. doi: 10.2106/00004623-199508000-00004. PMID 7642660
- [Background] Stein RB, Momose K, Bobet J. Biomechanics of human quadriceps muscles during electrical stimulation. J Biomech. 1999 Apr;32(4):347-57. doi: 10.1016/s0021-9290(98)00187-0. PMID 10213025
- [Background] Bruce-Brand RA, Walls RJ, Ong JC, Emerson BS, O'Byrne JM, Moyna NM. Effects of home-based resistance training and neuromuscular electrical stimulation in knee osteoarthritis: a randomized controlled trial. BMC Musculoskelet Disord. 2012 Jul 3;13:118. doi: 10.1186/1471-2474-13-118. PMID 22759883
- [Background] de Oliveira Melo M, Aragao FA, Vaz MA. Neuromuscular electrical stimulation for muscle strengthening in elderly with knee osteoarthritis - a systematic review. Complement Ther Clin Pract. 2013 Feb;19(1):27-31. doi: 10.1016/j.ctcp.2012.09.002. Epub 2012 Oct 18. PMID 23337561
- [Background] Vaz MA, Baroni BM, Geremia JM, Lanferdini FJ, Mayer A, Arampatzis A, Herzog W. Neuromuscular electrical stimulation (NMES) reduces structural and functional losses of quadriceps muscle and improves health status in patients with knee osteoarthritis. J Orthop Res. 2013 Apr;31(4):511-6. doi: 10.1002/jor.22264. Epub 2012 Nov 8. PMID 23138532
- [Background] Giggins O, Fullen B, Coughlan G. Neuromuscular electrical stimulation in the treatment of knee osteoarthritis: a systematic review and meta-analysis. Clin Rehabil. 2012 Oct;26(10):867-81. doi: 10.1177/0269215511431902. Epub 2012 Feb 9. PMID 22324059
- [Background] Osiri M, Welch V, Brosseau L, Shea B, McGowan J, Tugwell P, Wells G. Transcutaneous electrical nerve stimulation for knee osteoarthritis. Cochrane Database Syst Rev. 2000;(4):CD002823. doi: 10.1002/14651858.CD002823. PMID 11034768
- [Background] Mang CS, Clair JM, Collins DF. Neuromuscular electrical stimulation has a global effect on corticospinal excitability for leg muscles and a focused effect for hand muscles. Exp Brain Res. 2011 Mar;209(3):355-63. doi: 10.1007/s00221-011-2556-8. Epub 2011 Feb 1. PMID 21286692
- [Background] Dehail P, Duclos C, Barat M. Electrical stimulation and muscle strengthening. Ann Readapt Med Phys. 2008 Jul;51(6):441-51. doi: 10.1016/j.annrmp.2008.05.001. Epub 2008 Jun 18. English, French. PMID 18602713
- [Background] Paillard T. Combined application of neuromuscular electrical stimulation and voluntary muscular contractions. Sports Med. 2008;38(2):161-77. doi: 10.2165/00007256-200838020-00005. PMID 18201117
- [Background] Santos M, Zahner LH, McKiernan BJ, Mahnken JD, Quaney B. Neuromuscular electrical stimulation improves severe hand dysfunction for individuals with chronic stroke: a pilot study. J Neurol Phys Ther. 2006 Dec;30(4):175-83. doi: 10.1097/01.npt.0000281254.33045.e4. PMID 17233925
- [Background] Lagerquist O, Mang CS, Collins DF. Changes in spinal but not cortical excitability following combined electrical stimulation of the tibial nerve and voluntary plantar-flexion. Exp Brain Res. 2012 Oct;222(1-2):41-53. doi: 10.1007/s00221-012-3194-5. Epub 2012 Aug 17. PMID 22899312
- [Background] Shiba N, inventor. Kurume University, assignee. Apparatus for strengthening muscles. US patent 6,456,885. 2002 Sep 24.
- [Background] Yanagi T, Shiba N, Maeda T, Iwasa K, Umezu Y, Tagawa Y, Matsuo S, Nagata K, Yamamoto T, Basford JR. Agonist contractions against electrically stimulated antagonists. Arch Phys Med Rehabil. 2003 Jun;84(6):843-8. doi: 10.1016/s0003-9993(02)04948-1. PMID 12808536
- [Background] Mizusaki Imoto A, Peccin S, Gomes da Silva KN, de Paiva Teixeira LE, Abrahao MI, Fernandes Moca Trevisani V. Effects of neuromuscular electrical stimulation combined with exercises versus an exercise program on the pain and the function in patients with knee osteoarthritis: a randomized controlled trial. Biomed Res Int. 2013;2013:272018. doi: 10.1155/2013/272018. Epub 2013 Sep 14. PMID 24151589
- [Derived] Rabe KG, Matsuse H, Jackson A, Segal NA. Evaluation of the Combined Application of Neuromuscular Electrical Stimulation and Volitional Contractions on Thigh Muscle Strength, Knee Pain, and Physical Performance in Women at Risk for Knee Osteoarthritis: A Randomized Controlled Trial. PM R. 2018 Dec;10(12):1301-1310. doi: 10.1016/j.pmrj.2018.05.014. Epub 2018 May 29. PMID 29852286

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Intensity Exercise: 40% max isokinetic training in same repetitions/sets as experimental group.
  Isokinetic Training with Computer Sports Medicine Inc. (CSMi) HUMAC NORM: Low intensity exercises completed using CSMi HUMAC NORM in isokinetic mode at approximately 40%1 RM.
Period: Overall Study
Arm/Group | Hybrid Training | Low Intensity Exercise
Started | 21 | 21
Completed | 17 | 18
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hybrid Training | Low Intensity Exercise | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.62 (8.38) | 65.14 (9.51) | 66.38 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 165.38 (4.96) | 163.38 (8.53) | 164.4 (6.96)
Body Mass [Mean (Standard Deviation); unit: kilograms (kg)] | 74.49 (15.66) | 76.14 (15.56) | 75.31 (15.44)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.29 (5.99) | 28.45 (5.33) | 27.87 (5.64)
20-Meter Walk Time [Mean (Standard Deviation); unit: seconds] — A timed 20-meter walk was completed as a measure of lower limb physical performance. Participants were instructed to walk along a 20-meters straight, uninterrupted course as quickly as they could. Timing started when the participant initiated foot movement and stopped when both feet crossed the 20-meter mark. Times for two trials were recorded and the averaged.
  seconds | 13.12 (4.38) | 13.78 (3.22) | 13.49 (3.81)
5-Chair Stand Time [Mean (Standard Deviation); unit: seconds] — The chair stand test is a validated measure of physical performance in adults with knee osteoarthritis. Participants were instructed to stand from a chair (seat height 44.45 cm) 5 times as quickly as they could without using their arms. Two trials were timed and averaged.
  seconds | 17.13 (11.75) | 15.36 (4.35) | 16.25 (8.79)
Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain [Mean (Standard Deviation); unit: units on a scale] — The Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain subscale was used at baseline and follow-up to assess participant outcomes. The pain subscale is made up of 9 questions and was scored from zero to 100, with zero corresponding to extreme knee problems and 100 corresponding to no knee problems.
  units on a scale | 60.85 (15.47) | 54.86 (14.55) | 57.9 (15.07)
Extensor Torque [Mean (Standard Deviation); unit: Newton-meters] | 69.40 (3.67) | 67.60 (3.57) | 68.50 (3.62)
Flexor Torque [Mean (Standard Deviation); unit: Newton-meters] | 31.32 (1.82) | 28.36 (1.77) | 29.84 (1.80)

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximal Isokinetic Knee Extensor Torque by Body Mass Assessed by Isokinetic Dynamometer.
Description: Participants will be familiarized with strength testing equipment and counseled on proper lifting technique. They will undergo testing to determine their peak isokinetic knee extensor torque at 60°/sec, using an isokinetic dynamometer. These testing procedures will then be repeated for the other side.
Time Frame: Baseline and 12-week follow-up
Population: 4 participants in the hybrid training group discontinued the intervention due to unrelated pain, knee injections, car issues, and unrelated hospitalization. 3 participants in the low intensity exercise group discontinued the intervention due to unrelated pain, fatigue and the inability to gain strength due to radiation overdose (unrelated).
Measure: Least Squares Mean (Standard Error); unit: Newton-meters/kilogram
Groups:
- Low Intensity Exercise: Isokinetic Training with isokinetic dynamometer. Low intensity exercises completed in isokinetic mode at approximately 40%1 RM in same repetitions/sets as experimental group.
Arm/Group | Hybrid Training | Low Intensity Exercise
Number analyzed (Participants) | 17 | 18
Newton-meters/kilogram | 0.06 (0.04) | 0.03 (0.04)
Statistical Analysis 1: Comparison: Hybrid Training vs Low Intensity Exercise; Test type: Superiority; p = .67, Regression, Linear — Adjusted for two observations per subject; Side treated as a repeated factor

2. Secondary Outcome: Change in Maximal Isokinetic Knee Flexor Torque by Body Mass Assessed by Isokinetic Dynamometer.
Description: Participants will be familiarized with strength testing equipment and counseled on proper lifting technique. They will undergo testing to determine their peak isokinetic knee flexor torque, using an isokinetic dynamometer.
Time Frame: Baseline and 12-week follow-up
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Newton-meters/kilogram
Arm/Group | Hybrid Training | Low Intensity Exercise
Number analyzed (Participants) | 17 | 18
Newton-meters/kilogram | 0.05 (0.02) | 0.06 (0.02)

3. Secondary Outcome: Change in Knee Pain Assessed by a Knee Injury and Osteoarthritis Outcome Score
Description: The Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain subscale was used at baseline and follow-up to assess participant outcomes. The pain subscale is made up of 9 questions and was scored from zero to 100, with zero corresponding to extreme knee problems and 100 corresponding to no knee problems.
Time Frame: Baseline and 12-week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hybrid Training | Low Intensity Exercise
Number analyzed (Participants) | 17 | 18
units on a scale | 11.9 (11.5) | 14.1 (15.4)

4. Secondary Outcome: Change in 20-meter Walk Time
Description: A timed 20-meter walk was completed as a measure of lower limb physical performance. Participants were instructed to walk along a 20-meters straight, uninterrupted course as quickly as they could. Timing started when the participant initiated foot movement and stopped when both feet crossed the 20-meter mark. Times for two trials were recorded and the averaged.
Time Frame: Baseline and 12-week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Hybrid Training | Low Intensity Exercise
Number analyzed (Participants) | 17 | 18
seconds | -1.60 (2.04) | -0.95 (1.21)

5. Secondary Outcome: Change in 5-chair Stand Time
Description: The chair stand test is a validated measure of physical performance in adults with knee osteoarthritis. Participants were instructed to stand from a chair (seat height 44.45 cm) 5 times as quickly as they could without using their arms. Two trials were timed and averaged.
Time Frame: Baseline and 12-week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Hybrid Training | Low Intensity Exercise
Number analyzed (Participants) | 17 | 18
seconds | -4.81 (9.99) | -1.86 (4.72)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the duration of the study from baseline to 12-week follow-up.
Arm/Group | Hybrid Training | Low Intensity Exercise
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No